CLINICAL TRIAL: NCT02073552
Title: Randomized Clinical Trial to Evaluate the Colon Cleansing Quality of Polyethylene Glycol Compared With Polyethylene Glycol Plus Ascorbic Acid in Patients With Past Poor Colonic Preparation
Brief Title: Colon Cleansing Quality of Polyethylene Glycol Compared With Polyethylene Glycol Plus Ascorbic Acid.
Acronym: REPREP1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Responsible Party: Principal Investigator, Alberto Domínguez Rodríguez, MD,PhD, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REPREP1; 2013-002506-31 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2015-09

CONDITIONS: Colonoscopy Preparation
Keywords: colon cleansing, bowel preparations; polyethyleneglycol
MeSH Terms: interventions — polyethylene glycol 4000; polyethylene glycol 3350; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High volume (Active Comparator): * Two 5 mg bisacodyl tablets It is a stimulant laxative with local action.
  * Polyethylene glycol 4000: 16 envelopes (70 g of powder each). It includes electrolytes and sodium sulfate.
  Interventions: Drug: Polyethylene glycol 4000
- Low volume (Experimental): * Two 5 mg bisacodyl tablets, taken in the same way as for the high volume group.
  * Macrogol 3350 plus ascorbic acid: 4 envelopes, 2 containing 112 g polyethylene glycol and electrolytes and 2 with 2 g of ascorbic acid.
  Interventions: Drug: Macrogol 3350 plus ascorbic acid

INTERVENTIONS:
Drug: Polyethylene glycol 4000 — - Polyethylene glycol 4000: 16 envelopes (70 g of powder each). It includes electrolytes and sodium sulfate. These substances make PEG metabolically inert, achieving a suitable osmotic balance, despite having a high molecular weight. The preparation passes along the gastrointestinal tract without causing net absorption of fluid or electrolytes. It is routinely used in clinical practice for bowel cleansing, before abdominal surgery, barium enema and other colorectal and genitourinary tract tests. Participants will divide the whole doses in 4 liters of water taking half the day before the examination starting at 20.00 h and the other half at 6.00 pm on the day of the examination.
  Arms: High volume
Drug: Macrogol 3350 plus ascorbic acid — - Macrogol 3350 plus ascorbic acid: 4 envelopes, 2 containing 112 g polyethylene glycol and electrolytes and 2 with 2 g of ascorbic acid. The properties of the polyethylene glycol are the same as those mentioned previously, while ascorbic acid generates an osmotic gradient potentiating the effect of polyethylene glycol. It is used routinely as a bowel prep. Participants will divide the doses in 2 liters of water taking half the day before (112 g of PEG and an 11 g of ascorbic acid) the examination at 20.00 h and the other half at 6.00 pm on the day of the examination
  Arms: Low volume

SUMMARY:
The purpose of the study is to assess whether a low volume polyethylene glycol (PEG) plus ascorbic acid based bowel preparation for colonoscopy is not inferior to a large volume polyethylene glycol preparation in subjects with past history of poor bowel preparation

DETAILED DESCRIPTION:
Two key quality indicators for colonoscopy are the cecal intubation rate and the percentage of neoplastic lesions detected. Both factors are associated with adequate bowel cleansing. Poor cleansing ranged from 5% to 30% across studies, negatively affecting the efficiency of colonoscopy.

The most important factor associated with poor colonic preparation is the past history of poor bowel preparation. However, there are no recommendations on the proper type of preparation in those patients. In two non-randomized studies inadequate cleansing in the second colonoscopy ranged from 9.8% to 23%. Randomized studies comparing high volume (3-4 liters) with low volume (2 liters) PEG preparations, which are better tolerated by patients, are therefore needed before making any recommendations in this regard.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Outpatients with a history of past poor bowel prep, defined according to the Boston scale as a score less than 5.
* Signed informed consent

Exclusion Criteria:

paralytic ileus, intestinal obstruction, megacolon, poorly controlled hypertension (systolic pressure> 180, dyastolic pressure> 100), congestive heart failure, acute liver failure, end stage renal disease (dialysis or pre-dialysis), New York Heart Association class III-IV, pregnancy, diagnosis of phenylketonuria, diagnosis of glucose-6-phosphate dehydrogenase deficiency, dementia. History of poor preparation in the previous colonoscopy, colon resection, less than 75% intake of the bowel preparation in the index colonoscopy, refusal to participate in the study, patients in whom a new colonoscopy is not indicated despite a poor bowel preparation(i.e. ileal Crohn disease with poor large bowel preparation), lack of compliance with the bowel preparation schedule.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Colon cleansing | 30 days
  Colon cleansing will be assessed just after colonoscopy by the endoscopist in charge of performing the examination and afterwards images were reviewed by a the staff of endoscopists for validation (30 days). For assessing colon cleansing a validated scale (Boston scale) will be used.

SECONDARY OUTCOMES:
Tolerance of bowel preparation | Tolerance will be assessed just before colonoscopy by a research assistant
  It will be assessed by using a visual analog scale colon
Detection of colorectal neoplasia | 14 months
  Detection rate of adenoma and colorectal cancer will be assessed for both groups (low volume and high volume preparation)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z Gimeno García, MD, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Background] Atkin WS, Edwards R, Kralj-Hans I, Wooldrage K, Hart AR, Northover JM, Parkin DM, Wardle J, Duffy SW, Cuzick J; UK Flexible Sigmoidoscopy Trial Investigators. Once-only flexible sigmoidoscopy screening in prevention of colorectal cancer: a multicentre randomised controlled trial. Lancet. 2010 May 8;375(9726):1624-33. doi: 10.1016/S0140-6736(10)60551-X. Epub 2010 Apr 27. PMID 20430429
- [Background] Brenner H, Chang-Claude J, Jansen L, Knebel P, Stock C, Hoffmeister M. Reduced risk of colorectal cancer up to 10 years after screening, surveillance, or diagnostic colonoscopy. Gastroenterology. 2014 Mar;146(3):709-17. doi: 10.1053/j.gastro.2013.09.001. Epub 2013 Sep 5. PMID 24012982
- [Background] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM; ASGE/ACG Taskforce on Quality in Endoscopy. Quality indicators for colonoscopy. Am J Gastroenterol. 2006 Apr;101(4):873-85. doi: 10.1111/j.1572-0241.2006.00673.x. No abstract available. PMID 16635231
- [Background] Jover R, Herraiz M, Alarcon O, Brullet E, Bujanda L, Bustamante M, Campo R, Carreno R, Castells A, Cubiella J, Garcia-Iglesias P, Hervas AJ, Menchen P, Ono A, Panades A, Parra-Blanco A, Pellise M, Ponce M, Quintero E, Rene JM, Sanchez del Rio A, Seoane A, Serradesanferm A, Soriano Izquierdo A, Vazquez Sequeiros E; Spanish Society of Gastroenterology; Spanish Society of Gastrointestinal Endoscopy Working Group. Clinical practice guidelines: quality of colonoscopy in colorectal cancer screening. Endoscopy. 2012 Apr;44(4):444-51. doi: 10.1055/s-0032-1306690. Epub 2012 Mar 21. No abstract available. PMID 22438159
- [Background] ASGE Technology Committee; Mamula P, Adler DG, Conway JD, Diehl DL, Farraye FA, Kantsevoy SV, Kaul V, Kethu SR, Kwon RS, Rodriguez SA, Tierney WM. Colonoscopy preparation. Gastrointest Endosc. 2009 Jun;69(7):1201-9. doi: 10.1016/j.gie.2009.01.035. No abstract available. PMID 19481646
- [Background] Lorenzo-Zuniga V, Moreno-de-Vega V, Boix J. [Preparation for colonoscopy: types of scales and cleaning products]. Rev Esp Enferm Dig. 2012 Aug;104(8):426-31. doi: 10.4321/s1130-01082012000800006. Spanish. PMID 23039803
- [Background] Nyberg C, Hendel J, Nielsen OH. The safety of osmotically acting cathartics in colonic cleansing. Nat Rev Gastroenterol Hepatol. 2010 Oct;7(10):557-64. doi: 10.1038/nrgastro.2010.136. Epub 2010 Aug 24. PMID 20736921
- [Background] Chiu HM, Lin JT, Wang HP, Lee YC, Wu MS. The impact of colon preparation timing on colonoscopic detection of colorectal neoplasms--a prospective endoscopist-blinded randomized trial. Am J Gastroenterol. 2006 Dec;101(12):2719-25. doi: 10.1111/j.1572-0241.2006.00868.x. Epub 2006 Oct 6. PMID 17026559
- [Background] Parra-Blanco A, Nicolas-Perez D, Gimeno-Garcia A, Grosso B, Jimenez A, Ortega J, Quintero E. The timing of bowel preparation before colonoscopy determines the quality of cleansing, and is a significant factor contributing to the detection of flat lesions: a randomized study. World J Gastroenterol. 2006 Oct 14;12(38):6161-6. doi: 10.3748/wjg.v12.i38.6161. PMID 17036388
- [Background] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Background] Enestvedt BK, Tofani C, Laine LA, Tierney A, Fennerty MB. 4-Liter split-dose polyethylene glycol is superior to other bowel preparations, based on systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2012 Nov;10(11):1225-31. doi: 10.1016/j.cgh.2012.08.029. Epub 2012 Aug 30. PMID 22940741
- [Background] Corporaal S, Kleibeuker JH, Koornstra JJ. Low-volume PEG plus ascorbic acid versus high-volume PEG as bowel preparation for colonoscopy. Scand J Gastroenterol. 2010 Nov;45(11):1380-6. doi: 10.3109/00365521003734158. Epub 2010 Jul 5. PMID 20602568
- [Background] Ell C, Fischbach W, Bronisch HJ, Dertinger S, Layer P, Runzi M, Schneider T, Kachel G, Gruger J, Kollinger M, Nagell W, Goerg KJ, Wanitschke R, Gruss HJ. Randomized trial of low-volume PEG solution versus standard PEG + electrolytes for bowel cleansing before colonoscopy. Am J Gastroenterol. 2008 Apr;103(4):883-93. doi: 10.1111/j.1572-0241.2007.01708.x. Epub 2008 Jan 11. PMID 18190651
- [Background] Gentile M, De Rosa M, Cestaro G, Forestieri P. 2 L PEG plus ascorbic acid versus 4 L PEG plus simethicon for colonoscopy preparation: a randomized single-blind clinical trial. Surg Laparosc Endosc Percutan Tech. 2013 Jun;23(3):276-80. doi: 10.1097/SLE.0b013e31828e389d. PMID 23751992
- [Background] Marmo R, Rotondano G, Riccio G, Marone A, Bianco MA, Stroppa I, Caruso A, Pandolfo N, Sansone S, Gregorio E, D'Alvano G, Procaccio N, Capo P, Marmo C, Cipolletta L. Effective bowel cleansing before colonoscopy: a randomized study of split-dosage versus non-split dosage regimens of high-volume versus low-volume polyethylene glycol solutions. Gastrointest Endosc. 2010 Aug;72(2):313-20. doi: 10.1016/j.gie.2010.02.048. Epub 2010 Jun 19. PMID 20561621
- [Background] Pontone S, Angelini R, Standoli M, Patrizi G, Culasso F, Pontone P, Redler A. Low-volume plus ascorbic acid vs high-volume plus simethicone bowel preparation before colonoscopy. World J Gastroenterol. 2011 Nov 14;17(42):4689-95. doi: 10.3748/wjg.v17.i42.4689. PMID 22180711
- [Background] Jansen SV, Goedhard JG, Winkens B, van Deursen CT. Preparation before colonoscopy: a randomized controlled trial comparing different regimes. Eur J Gastroenterol Hepatol. 2011 Oct;23(10):897-902. doi: 10.1097/MEG.0b013e32834a3444. PMID 21900786
- [Background] Lebwohl B, Wang TC, Neugut AI. Socioeconomic and other predictors of colonoscopy preparation quality. Dig Dis Sci. 2010 Jul;55(7):2014-20. doi: 10.1007/s10620-009-1079-7. Epub 2010 Jan 16. PMID 20082217
- [Background] Ness RM, Manam R, Hoen H, Chalasani N. Predictors of inadequate bowel preparation for colonoscopy. Am J Gastroenterol. 2001 Jun;96(6):1797-802. doi: 10.1111/j.1572-0241.2001.03874.x. PMID 11419832
- [Background] Ben-Horin S, Bar-Meir S, Avidan B. The outcome of a second preparation for colonoscopy after preparation failure in the first procedure. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):626-30. doi: 10.1016/j.gie.2008.08.027. PMID 19251002
- [Background] Ibanez M, Parra-Blanco A, Zaballa P, Jimenez A, Fernandez-Velazquez R, Fernandez-Sordo JO, Gonzalez-Bernardo O, Rodrigo L. Usefulness of an intensive bowel cleansing strategy for repeat colonoscopy after preparation failure. Dis Colon Rectum. 2011 Dec;54(12):1578-84. doi: 10.1097/DCR.0b013e31823434c8. PMID 22067188
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Derived] Gimeno-Garcia AZ, Hernandez G, Aldea A, Nicolas-Perez D, Jimenez A, Carrillo M, Felipe V, Alarcon-Fernandez O, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Moreno M, Ramos L, Quintero E. Comparison of Two Intensive Bowel Cleansing Regimens in Patients With Previous Poor Bowel Preparation: A Randomized Controlled Study. Am J Gastroenterol. 2017 Jun;112(6):951-958. doi: 10.1038/ajg.2017.53. Epub 2017 Mar 14. PMID 28291237